CLINICAL TRIAL: NCT03335488
Title: A Randomised, Controlled, Open-Label Parallel Arm Study of Safety, PK and Ammonia Control of RAVICTI® (Glycerol Phenylbutyrate) Oral Liquid and Sodium Phenylbutyrate in Phenylbutyrate Treatment Naïve Patients With Urea Cycle Disorders
Brief Title: Study of Glycerol Phenylbutyrate & Sodium Phenylbutyrate in Phenylbutyrate Naïve Patients With Urea Cycle Disorders (UCDs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPN-100-021; 2015-000075-27 (EudraCT Number)
Record Dates: First submitted 2017-10-18; First posted 2017-11-07 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorder
Keywords: Urea; Hyperammonemic crisis (HAC)
MeSH Terms: conditions — Urea Cycle Disorders, Inborn | interventions — glycerol phenylbutyrate; 4-phenylbutyric acid

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled, Open-Label Parallel Arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RAVICTI -> RAVICTI (Experimental): Initial Treatment, Maintenance, Safety Extension Periods: RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose. Dosing will be based on participants disease and treatment status at entry to the study.
  Interventions: Drug: RAVICTI
- NaPBA -> RAVICTI (Active Comparator): Initial Treatment Period: NaPBA dosing based on participants disease and treatment status at entry to the study.
  Transition, Maintenance, Safety Extension Periods: RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose. Dosing will be based on participants disease and treatment status at entry to the study.
  Interventions: Drug: NaPBA

INTERVENTIONS:
Drug: RAVICTI — RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose
  Other Names: Glycerol phenylbutyrate; GPB; HPN-100
  Arms: RAVICTI -> RAVICTI
Drug: NaPBA — * NaPBA in patients weighing < 20 Kg - 600 mg/Kg, maximum total daily dose
  * NaPBA in patients weighing > 20 Kg - 13 g/m2, maximum total daily dose
  Other Names: Sodium phenylbutyrate
  Arms: NaPBA -> RAVICTI

SUMMARY:
This is a randomized, controlled, open-label parallel arm study to assess the safety, tolerability, pharmacokinetics and ammonia control, of RAVICTI® as compared to Sodium phenylbutyrate (NaPBA) in urea cycle disorder subjects not currently or previously chronically treated with phenylacetic acid (phenylacetate; PAA) prodrugs. The study design will include: 1) Baseline Period; 2) Initial Treatment Period; 3) a RAVICTI only Transition Period 4) a RAVICTI only Maintenance Period; and 5) a RAVICTI only Safety Extension Period. The study will run for approximately 25 weeks.

DETAILED DESCRIPTION:
Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent given by the subject or the subject's parent/legal guardian for those under 18 years of age or the age of consent by local regulation.
* Male and female subjects with a suspected or confirmed UCD diagnosis of any subtype, except n-acetylglutamate synthetase (NAGS) deficiency.
* Suspected diagnosis is defined as having experienced a hyperammonemic crisis (HAC) or a documented high ammonia of >=100 µmol/L
* Confirmed diagnosis is determined via enzymatic, biochemical, or genetic testing.

  * Requires nitrogen-binding agents according to the judgment of the Investigator
  * Birth and older.
  * All females of childbearing potential and all sexually active males must agree to use an acceptable method of contraception from signing the informed consent throughout the study and for 30 days after the last dose of study drug. Acceptable forms of contraception are (oral, injected, implanted or transdermal), tubal ligation, intrauterine device, hysterectomy, vasectomy, or double barrier methods. Abstinence is an acceptable form of birth control, though appropriate contraception must be used if the subject becomes sexually active.

Exclusion Criteria:

* Subject has received chronic treatment with an oral phenylbutyrate (RAVICTI, NaPBA, Pheburane, or other) longer than 14 consecutive days within one year prior to enrollment.
* Temporary use of NaPBA for acute management of a hyperammonemic crisis in the past is acceptable.

  * Any concomitant illness (e.g., malabsorption or clinically significant liver or bowel disease) which would preclude the subject's safe participation, as judged by the Investigator.
  * Has undergone liver transplantation, including hepatocellular transplant.
  * Subjects on sodium benzoate (NaBz) at Baseline will be excluded if they are viewed by the Investigator as being unable to undergo NaBz transition to a PAA prodrug during the Initial Treatment Period.
  * Known hypersensitivity to phenylbutyric acid (PBA) or any excipients of the NaPBA/PBA formulations.
  * Pregnant or breast-feeding patients. Women of childbearing potential must have a pregnancy test performed at the Baseline Visit prior to the start of study drug.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (6):
  - University of Florida (UF) - Shands Hospital, Gainesville, Florida
  - Mount Sinai School of Medicine, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Texas, Southwestern Medical Centre, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- Italy (2):
  - Azienda Ospedaliera Universitaria Di Padova, U.O.C. Malattie Metaboliche Ereditarie, Dipartimento della Salute della Donna e del Bambino, Padua, Veneto
  - Bambino Gesù Children's Research Hospital, Rome
- Spain (2):
  - Hospital Materno-Infantil (HRU Carlos Haya), Málaga, Andalusia
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
- Universitätsspital, Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Initial Treatment Period (approximately 28 days), eligible participants were randomized to one of two treatment arms: RAVICTI or NaPBA. For all Initial Treatment Period NaPBA participants and RAVICTI participants who were treatment failures, a Transition Period (7 days ± 2 days) with RAVICTI followed. All participants received RAVICTI in the Maintenance Period (8 Weeks) and the Safety Extension Period (12 Weeks).
Groups:
- NaPBA -> RAVICTI: Initial Treatment Period: NaPBA dosing based on participants disease and treatment status at entry to the study:
  * NaPBA in patients weighing < 20 Kg - 600 mg/Kg, maximum total daily dose
  * NaPBA in patients weighing > 20 Kg - 13 g/m2, maximum total daily dose.
  Transition, Maintenance, Safety Extension Periods: RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose. Dosing will be based on participants disease and treatment status at entry to the study.
Period: Initial Treatment Period
Arm/Group | RAVICTI -> RAVICTI | NaPBA -> RAVICTI
Started | 11 | 5
Completed | 11 | 5
Not Completed | 0 | 0
Period: Transition Period
Arm/Group | RAVICTI -> RAVICTI | NaPBA -> RAVICTI
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0
Period: Maintenance Period
Arm/Group | RAVICTI -> RAVICTI | NaPBA -> RAVICTI
Started | 11 | 5
Completed | 10 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0
Period: Safety Extension Period
Arm/Group | RAVICTI -> RAVICTI | NaPBA -> RAVICTI
Started | 10 | 5
Completed | 8 | 5
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Did Not Return to Study Visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- NaPBA -> RAVICTI: Initial Treatment Period: NaPBA dosing based on participants disease and treatment status at entry to the study:
  NaPBA in patients weighing < 20 Kg - 600 mg/Kg, maximum total daily dose NaPBA in patients weighing > 20 Kg - 13 g/m2, maximum total daily dose.
  Transition, Maintenance, Safety Extension Periods: RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose. Dosing will be based on participants disease and treatment status at entry to the study.
- Total: Total of all reporting groups
Arm/Group | RAVICTI -> RAVICTI | NaPBA -> RAVICTI | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Customized [Count of Participants; unit: Participants]
  < 2 months | 1 | 0 | 1
  2 months - < 2 years | 4 | 0 | 4
  2 years - 12 years | 1 | 3 | 4
  > 12 - 16 years | 0 | 0 | 0
  >= 17 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 5 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Treatment Success (Percentage of Participants Defined as Treatment Success at Week 4) During the Initial Treatment Period
Description: A participant was considered a Treatment Success for the assigned treatment arm if the participant had not experienced an unprovoked hyperammonemic crisis (HAC) (i.e., a HAC that cannot be attributed to one or more specific precipitating factors such as infection, intercurrent illness, diet noncompliance, treatment noncompliance, etc.) on the assigned treatment and had met at least 2 of the following 3 criteria:
  * Had absolute values at the 3 time points (pre-dose, after dose at 4 hours and 8 hours) of plasma ammonia levels which do not exceed ULN at the Week 4(End of Initial Treatment Period visit)
  * Had normal (≤ ULN) glutamine levels at the Week 4 (End of Initial Treatment Period visit at the time point Zero Hour.
  * Had normal (≤ ULN) essential amino acids including branched chain amino acid levels (threonine, phenylalanine, methionine, lysine, leucine, isoleucine, histidine, valine) at the End of Initial Treatment Period visit at time point Zero Hour.
Time Frame: Week 4
Population: Modified Intent-to-Treat Population: all participants from the Safety population with no major eligibility violations and participants who had ammonia data post-randomization.
Measure: Number; unit: percentage of participants
Groups:
- RAVICTI: Initial Treatment Period: RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose. Dosing will be based on participants disease and treatment status at entry to the study.
- NaPBA: Initial Treatment Period: NaPBA dosing based on participants disease and treatment status at entry to the study:
  NaPBA in patients weighing < 20 Kg - 600 mg/Kg, maximum total daily dose NaPBA in patients weighing > 20 Kg - 13 g/m2, maximum total daily dose.
Arm/Group | RAVICTI | NaPBA
Number analyzed (Participants) | 11 | 5
percentage of participants | 81.8 | 80.0
Statistical Analysis 1: Comparison: RAVICTI vs NaPBA; Test type: Superiority; p = 1.0000, Fisher Exact; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.0 to 28.1]

2. Secondary Outcome: Rate of Drug Discontinuations (Percentage of Participants Who Discontinued Study Drug) Due to Any Reason in the Initial Treatment Period
Time Frame: Baseline through Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | RAVICTI | NaPBA
Number analyzed (Participants) | 11 | 5
percentage of participants | 0 | 0

3. Secondary Outcome: Change From Baseline in Fasting Plasma Ammonia Levels During the Initial Treatment Period
Time Frame: Baseline, Initial Treatment Period Week 1, Week 2, Week 3, Week 4 (0, 4, 8 hours post dose)
Population: Modified Intent-to-Treat Population: all participants from the Safety population with no major eligibility violations and participants who had ammonia data post-randomization. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RAVICTI | NaPBA
Number analyzed (Participants) | 11 | 5
µmol/L
  Week 1 | 6.5 (21.16) | 0.0 (10.12)
  Week 2: number analyzed (Participants) | 11 | 4
  Week 2 | 25.5 (59.88) | -10.4 (10.17)
  Week 3: number analyzed (Participants) | 10 | 4
  Week 3 | 7.4 (35.91) | -10.9 (6.40)
  Week 4: 0 hour | 2.1 (15.52) | -0.3 (8.49)
  Week 4: 4 hours postdose: number analyzed (Participants) | 8 | 5
  Week 4: 4 hours postdose | 2.6 (23.49) | -1.1 (8.68)
  Week 4: 8 hours postdose: number analyzed (Participants) | 10 | 5
  Week 4: 8 hours postdose | 23.4 (62.09) | -0.7 (7.37)
Statistical Analysis 1: Comparison: RAVICTI vs NaPBA; Initial Treatment Period Week 1; Test type: Superiority; p = 0.8464, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: RAVICTI vs NaPBA; Initial Treatment Period Week 2; Test type: Superiority; p = 0.1040, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: RAVICTI vs NaPBA; Initial Treatment Period Week 3; Test type: Superiority; p = 0.0979, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: RAVICTI vs NaPBA; End of Initial Treatment Period Week 4 - 0 Hr; Test type: Superiority; p = 0.9808, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: RAVICTI vs NaPBA; End of Initial Treatment Period Week 4 - 4 Hr; Test type: Superiority; p = 0.8329, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: RAVICTI vs NaPBA; End of Initial Treatment Period Week 4 - 8 Hr; Test type: Superiority; p = 0.2544, Wilcoxon rank sum test

4. Secondary Outcome: Plasma Ammonia Area Under the Curve (AUC) 0 to 8h at the End of the Initial Treatment Period
Time Frame: Week 4: hour 0 (predose), and hours 4 and 8 postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µmol*h /L
Arm/Group | RAVICTI | NaPBA
Number analyzed (Participants) | 10 | 5
µmol*h /L | 331.8 (342.79) | 258.9 (153.35)
Statistical Analysis 1: Comparison: RAVICTI vs NaPBA; Test type: Superiority; p = 0.8579, t-test — P-value is from a t-test comparing log-transformed RAVICTI vs NaPBA values

5. Secondary Outcome: Peak Plasma Concentration (Cmax) of Ammonia at the End of the Initial Treatment Period
Time Frame: Week 4: hour 0 (predose), and hours 4 and 8 postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RAVICTI | NaPBA
Number analyzed (Participants) | 11 | 5
µmol/L | 60.2 (78.47) | 38.1 (18.91)
Statistical Analysis 1: Comparison: RAVICTI vs NaPBA; Test type: Superiority; p = 0.7155, t-test — P-value is from a t-test comparing log-transformed RAVICTI vs NaPBA values

ADVERSE EVENTS:
Time Frame: All-cause mortality: from enrollment through the end of study up to 25 weeks plus 30 days. Adverse events: from the first dose through the last dose of study drug in a given period, plus 30 days from the last dose taken, regardless of period. Overall mean time on treatment for the Initial Treatment Period was 30.7 days (RAVICTI) and 26.0 days (NaPBA), for the Transition Period was 8.0 days, for the Maintenance Period was 54.4 days, and for the Safety Extension Period was 84.6 days.
Groups:
- Initial Treatment Period: RAVICTI: RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose for up to 28 days.
- Initial Treatment Period: NaPBA: Initial Treatment Period: NaPBA for up to 28 days dosing based on participants disease and treatment status at entry to the study:
  NaPBA in patients weighing < 20 Kg - 600 mg/Kg, maximum total daily dose NaPBA in patients weighing > 20 Kg - 13 g/m2, maximum total daily dose.
- Transition Period: RAVICTI: RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose for 7 days ± 2 days
- Maintenance and Safety Periods Combined: RAVICTI, Oral Liquid Product 17.5 mL maximum total daily dose in the Maintenance Period (8 Weeks) and the Safety Extension Period (12 Weeks)
Arm/Group | Initial Treatment Period: RAVICTI | Initial Treatment Period: NaPBA | Transition Period: RAVICTI | Maintenance and Safety Periods Combined
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/5 | 0/5 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/5 | 1/5 | 3/16
Other Adverse Events (participants affected / at risk) | 6/11 | 2/5 | 1/5 | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Period: RAVICTI (N=11) | Initial Treatment Period: NaPBA (N=5) | Transition Period: RAVICTI (N=5) | Maintenance and Safety Periods Combined (N=16)
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperammonaemic crisis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment Period: RAVICTI (N=11) | Initial Treatment Period: NaPBA (N=5) | Transition Period: RAVICTI (N=5) | Maintenance and Safety Periods Combined (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Amino acid level decreased (Investigations) | 1 | 0 | 0 | 0
Ammonia increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT03335488/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03335488/SAP_001.pdf